CLINICAL TRIAL: NCT07273370
Title: A Study on Child Speech Data Collection for a Diagnostic App Targeting Delayed Articulation in Children
Brief Title: Child Speech Data Collection
Status: Completed | Type: Observational
Sponsor: JeeHyun Suh (Other)
Collaborators: National IT Industry Promotion Agency, Republic of Korea (Unknown)
Responsible Party: Sponsor-Investigator, JeeHyun Suh, PI, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Other Study IDs: B-2510-1000-306
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Children; Developmental Delays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children: 2~13 years of children
  Interventions: Diagnostic Test: U-TAP; Diagnostic Test: hidongdong

INTERVENTIONS:
Diagnostic Test: U-TAP — A Korean-based language/articulation development assessment that evaluates consonant accuracy, vowel accuracy, and other aspects by having the subject pronounce listed words.
Diagnostic Test: hidongdong — This is a Korean-based language/pronunciation development assessment newly developed using the Delphi methodology for digital transformation. It evaluates consonant accuracy, vowel accuracy, and other aspects by having subjects pronounce presented words.

SUMMARY:
Verify the non-inferiority of Korea's language development assessment U-TAP and the self-developed language development assessment 'Hi Dongdong', and verify the non-inferiority of speech-language pathologist-based assessment versus AI-based assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2 to under 14 years old
2. Children possessing cognitive abilities sufficient to understand basic instructions and follow simple directions
3. Cases where the child's guardian has received a thorough explanation of the research purpose, methods, personal information, and voice data processing policies, and has signed the research consent form
4. Individuals who understand and consent to the research purpose and survey methods
5. Individuals meeting all criteria listed in the above selection criteria

Exclusion Criteria:

1. Cases where guardian consent has not been secured
2. Cases where consent has not been obtained for the Personal Information and Voice Data Usage Agreement
3. Children unable to perform research tasks due to moderate or higher intellectual disability
4. Children with temporarily distorted voice characteristics due to acute illness (e.g., respiratory disease)
5. When the recording environment (maintaining concentration, prompting speech) cannot be secured
6. When any of the criteria listed in the above exclusion criteria apply

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: korean(south)
Sampling Method: Non-Probability Sample
Enrollment: 931 (Actual)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
U-TAP | baseline
  Urimal Test of Articulation and Phonology
hi-dongdong | Day 1
  Newly developed language assessment tool

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided